CLINICAL TRIAL: NCT02589444
Title: Pilot Study Evaluating the Role of Vitamin D Repletion on Gut and Lung Microbiota in Cystic Fibrosis
Brief Title: Vitamin D and Microbiota in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, MD, PH.D, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00083796
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Vitamin D Deficiency; Cystic Fibrosis
Keywords: Clinical Endocrinology; Immunology; Inflammation; Microbiology; Respiratory Disorders; Vitamins
MeSH Terms: conditions — Vitamin D Deficiency; Cystic Fibrosis; Inflammation; Respiration Disorders | interventions — Cholecalciferol; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Participants with vitamin D deficiency - treatment group (Experimental): Participants with 25-hydroxyvitamin D (25(OH)D) ≤30 ng/mL taking oral high-dose vitamin D3 (50,000 IU) once a week and providing stool and sputum sample at screening and 3 months after screening.
  Interventions: Dietary Supplement: High-Dose Vitamin D3; Other: Stool Sample; Other: Sputum Sample; Procedure: Blood draw
- Participants with vitamin D deficiency - placebo group (Sham Comparator): Participants with 25-hydroxyvitamin D (25(OH)D) concentrations ≤30 ng/mL taking a sham comparator (placebo) once a week and providing stool sample and sputum sample at screening and 3 months after screening.
  Interventions: Other: Stool Sample; Other: Sputum Sample; Other: Sham Comparator; Procedure: Blood draw
- Participants without vitamin D deficiency (Other): Participants with 25-hydroxyvitamin D (25(OH)D) concentrations > 30 ng/mL with no intervention and providing stool sample and sputum sample at screening and 3 months after screening.
  Interventions: Other: Stool Sample; Other: Sputum Sample; Procedure: Blood draw

INTERVENTIONS:
Dietary Supplement: High-Dose Vitamin D3 — 50,000 IU of oral vitamin D3 once a week (the standard of care for repletion of vitamin D status by the Cystic fibrosis Foundation)
  Other Names: Cholecalciferol
  Arms: Participants with vitamin D deficiency - treatment group
Other: Stool Sample — Participants will be asked to provide a stool sample in a collection container for analysis of stool microbiota. This will be done upon enrollment (baseline) and at 3 month follow-up.
Other: Sputum Sample — Participants will be asked to collect their sputum (the thick mucus or phlegm that is expelled from the lower respiratory tract through coughing) into a kit.
  This will be done upon enrollment (baseline) and at 3 month follow-up.
Other: Sham Comparator — A placebo capsule taken once a week (manufactured by the same company that makes the Vitamin D supplement).
  Other Names: Placebo
  Arms: Participants with vitamin D deficiency - placebo group
Procedure: Blood draw — Participants will be asked to provide 30 ml of blood collected via a blood draw to measure 25 (OH)D serum concentration and other nutrient markers related to vitamin D including Parathyroid hormone, fibroblast growth factor-23, vitamin D binding protein and markers of immune system/inflammation. This will be done at baseline and at 3 months follow up.

SUMMARY:
The objective of this study is to assess the effects of a high-dose vitamin D3 on the composition of gut and lung microbiota in adolescents and adults with cystic fibrosis who are vitamin D deficient.

DETAILED DESCRIPTION:
Monocentric, double-blind, randomized, placebo-controlled, interventional pilot study to investigate the beneficial effects of high dose vitamin D supplementation on gut and lung microbiota in patients with cystic fibrosis who are vitamin D insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the Cystic fibrosis clinic for routine follow up of cystic fibrosis
* Serum 25(OH)D concentrations obtained within 2 months of enrollment
* Able to tolerate oral medications

Exclusion Criteria:

* Inability to obtain or declined informed consent from the subject and/or legally authorized representative
* Pregnancy or plans to become pregnant in the next 3 months
* History of disorders associated with hypercalcemia including parathyroid disease
* Current hypercalcemia (albumin-corrected serum calcium >10.8 mg/dL or ionized calcium >5.2 mg/dL)
* History of nephrolithiasis with active symptoms within the past two years
* Chronic kidney disease worse than stage III (<60 ml/min)
* Current significant hepatic dysfunction total bilirubin > 2.5 mg/dL with direct bilirubin > 1.0 mg/dL
* Current use of cytotoxic or immunosuppressive drugs
* History of AIDS
* History of illicit drug abuse (defined as history of enrollment into a drug rehabilitation program or hospital visits due to drug use within the past 3 years or any use of the following drugs in the past 6 months (cocaine, opiates, amphetamines, marijuana) or any positive toxicology screen for (cocaine, opiates, amphetamines, marijuana)
* Too ill to participate in study based on investigator's or study team's opinion
* Current enrollment in another intervention trial
* In addition we amended our study with three additional criteria 11) systemic antibiotic use in the last 4 weeks, 12) use of probiotics and, 13) inflammatory bowel disease, four months after the start of the study and after 12 subjects were randomized, as we considered that these factors may also influence our study endpoints. Of the 12 subjects who were randomized, only 4 would have been excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Shannon Index | Change from baseline shannon Index at 3 months after initiation of treatment
  Sputum microbiota analysis will be measured using this ecological diversity measure. Sputum samples will be collected via a sputum kit.
Species Richness Index | Change from baseline Species Richness Index at 3 months after initiation of treatment
  Stool microbiota analysis will be measured using this ecological diversity measure. Stool samples will be collected using a stool kit provided to the participant.

SECONDARY OUTCOMES:
Serum 25(OH)D levels (and other nutritional markers related to vitamin D including nutrient levels, parathyroid hormone, fibroblast growth factor-23, free 25(OH)D, vitamin D binding protein | At baseline and 3 months after initiation of treatment
  Collected via blood draw.
Forced expiratory volume in 1 second (FEV1) | Change in Forced expiratory volume in 1 second( FEV1) at 3 months after initiation of treatment
  Spirometry (is a common office test used to assess how well the participant's lungs work by measuring how much air the participant inhales, how much the participant exhales and how quickly the participant exhales) to assess the impact of vitamin D status on lung function.
  Spirometry results will only be collected if they are done as part of the participants routine care.
Measures of plasma oxidative stress by assessing plasma aminothiol concentrations (glutathione, glutathione disulfide, cysteine, cystine) and their redox potentials. | At baseline and 3 months after initiation of treatment
  Collected via blood draw.
Measures of inflammation by assessing plasma IL-6, TNF-alpha, MCP-1, and IL-8 concentrations | At baseline and 3 months after initiation of treatment
  Collected via blood draw.
Forced vital capacity (FVC) | Change in Forced vital capacity( FVC) at 3 months after initiation of treatment
  Spirometry (is a common office test used to assess how well the participant's lungs work by measuring how much air the participant inhales, how much the participant exhales and how quickly the participant exhales) to assess the impact of vitamin D status on lung function.
  Spirometry results will only be collected if they are done as part of the participants routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD/PhD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Kanhere M, He J, Chassaing B, Ziegler TR, Alvarez JA, Ivie EA, Hao L, Hanfelt J, Gewirtz AT, Tangpricha V. Bolus Weekly Vitamin D3 Supplementation Impacts Gut and Airway Microbiota in Adults With Cystic Fibrosis: A Double-Blind, Randomized, Placebo-Controlled Clinical Trial. J Clin Endocrinol Metab. 2018 Feb 1;103(2):564-574. doi: 10.1210/jc.2017-01983. PMID 29161417